CLINICAL TRIAL: NCT05977998
Title: A Phase II Study of Perioperative Paclitaxel in Patients With Gastric Adenocarcinoma and Carcinomatosis or Positive Cytology
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0331; NCI-2023-05915 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-07-24; First posted 2023-08-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Gastric Adenocarcinoma; Carcinomatosis
MeSH Terms: conditions — Carcinoma | interventions — Paclitaxel; Dexamethasone; Calcium Dobesilate; Diphenhydramine; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Paclitaxel (Experimental): Participant will receive paclitaxel every 2 weeks for 6 weeks, and then participants may have a gastrectomy based on what the doctor thinks is in your best interest. You may then receive additional paclitaxel every 2 weeks for 6 weeks.
  Interventions: Drug: Paclitaxel; Drug: Dexamethasone; Drug: Diphenhydramine; Drug: Famotidine

INTERVENTIONS:
Drug: Paclitaxel — Given by IP (Intraperitoneal injection)
  Other Names: Taxol
Drug: Dexamethasone — Given by IV (vein)
  Other Names: Decadron
Drug: Diphenhydramine — Given by IV (vein)
  Other Names: Benadryl®
Drug: Famotidine — Given by IV (vein)
  Other Names: Pepcid®

SUMMARY:
To learn about the effects of paclitaxel and gastrectomy (surgery to remove all or part of the stomach) on improving outcomes in patients with gastric cancer.

DETAILED DESCRIPTION:
Primary Objectives:

To assess overall survival from the date of diagnosis in subjects with stage IV gastric or gastroesophageal cancer and positive cytology or carcinomatosis after perioperative intraperitoneal paclitaxel and gastrectomy.

Secondary Objectives:

To assess the safety of gastrectomy in subjects with stage IV gastric or gastroesophageal cancer and positive cytology or carcinomatosis undergoing treatment with perioperative intraperitoneal paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above. There will be no upper age restriction. Because no dosing or adverse event data are currently available on the use of intraperitoneal paclitaxel in patients <18 years of age, children are excluded from this study.
2. ECOG performance status ≤ 2 (Karnofsky ≥60%). Appendices 1 and 2.
3. Cytologic or histologic proof of adenocarcinoma of the stomach or gastroesophageal junction.
4. Adequate renal, and bone marrow function:

   1. Leukocytes >= 3,000/uL
   2. Absolute neutrophil count >= 1,500/uL
   3. Platelets >= 60,000/Ul
   4. Serum creatinine <= 1.6 mg/dL
5. Distant Metastatic Disease of peritoneum:

   1. Positive peritoneal cytology, or
   2. Carcinomatosis on diagnostic laparoscopy or laparotomy.
6. Completion of preoperative systemic cytotoxic chemotherapy. Targeted therapy, such as HER2 directed therapy, and immunotherapy, such as PD-1 inhibitors, may be continued.
7. English and non-English speaking patients are eligible.

Exclusion Criteria:

1. Distant metastatic disease not limited to the peritoneum such as solid organ metastases to the liver, central nervous system, or lung.
2. Infections such as pneumonia or wound infections that would preclude protocol therapy.
3. Women with a positive urine or serum pregnancy test are excluded from this study; women of childbearing potential (defined as those who are not postmenopausal defined as no menses in greater than or equal to 12 months, have not had a hysterectomy or bilateral salpingo-oophorectomy, do not have ovarian failure, or have not had a surgical sterilization procedure) must agree to refrain from breast-feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, a double barrier method, or abstinence. Men with reproductive potential must agree to an appropriate method of birth control, including abstinence or double barrier method (diaphragm plus condom).
4. Subjects with unstable angina or New York Heart Association Grade II or greater congestive heart failure.
5. Subjects, such as those with cognitive impairment, deemed unable to comply with study and/or follow-up procedures.
6. Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity.
7. Previous surgery that would preclude safe cytoreduction and intraperitoneal port placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Badgwell, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT05977998/ICF_000.pdf